CLINICAL TRIAL: NCT04943991
Title: Fabry Disease in High-risk Patients With Left Ventricular Hypertrophy: Prevalence and Implementation of a Clinical Score
Acronym: FAPREV-HCM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FAPREV-HCM
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Fabry Disease; Fabry Disease, Cardiac Variant; Lysosomal Storage Diseases; HCM - Hypertrophic Cardiomyopathy; Anderson Fabry Disease
Keywords: prevalence; fabry disease; HCM; hypertrophic cardiomyopathy; rare disease; diagnostics; lysosomal storage diseasese
MeSH Terms: conditions — Fabry Disease; Fabry Disease, Cardiac Variant; Lysosomal Storage Diseases; Cardiomyopathy, Hypertrophic; Rare Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HCM/LVH at University Hospital Wuerzburg (Other)
  Interventions: Diagnostic Test: blood sampling (alpha-Galactosidase & LysoGb3)

INTERVENTIONS:
Diagnostic Test: blood sampling (alpha-Galactosidase & LysoGb3) — A blood sample will be taken. Alpha-Galactosidase level and LysoGb3 will be measured.
  Amendment: Offering of genetic testing for fabry specific GLA-gene

SUMMARY:
This study aims to evaluate the prevalence of Fabry Disease (FD) among a cohort of high risk patients with left ventricular hypertrophy (LVH) presenting at the University Hospital Würzburg over the last 20 years. Fabry disease is a rare disease that is known to be consistently underdiagnosed due to its largely variable symptoms.

Considering that an early Fabry diagnosis is crucial for maximum benefit from therapies available, screening for Fabry patients can contribute to preventing development and worsening of symptoms in Fabry patients with LVH.

In addition, a positive diagnosis in a family member opens the possibility to diagnose further family members in an earlier stage of the disease, therefore allowing treatment of symptoms and organ manifestations before they become irreversible.

DETAILED DESCRIPTION:
Aims of the study:

To evaluate the prevalence of Fabry Disease (FD) among a cohort of high risk patients with left ventricular hypertrophy (LVH) presenting at the University Hospital Würzburg over the last 10 years. Fabry disease is a rare disease that is known to be consistently underdiagnosed due to its largely variable symptoms. Considering that an early Fabry diagnosis is crucial for maximum benefit from therapies available, screening for Fabry patients can contribute to preventing development and worsening of symptoms in Fabry patients with LVH. In addition, a positive diagnosis in a family member opens the possibility to diagnose further family members in an earlier stage of the disease, therefore allowing treatment of symptoms and organ manifestations before they become irreversible.

Background:

Fabry disease (FD) is a rare X-linked disease caused by enzyme α-Galactosidase A (αGAL) deficiency resulting from mutations in the gene encoding this enzyme. Many patients present with a "private" specific mutation found only in that particular family and, thus, several hundreds of mutations are currently known. This multiplicity in mutations contributes to large variations in residual enzyme activity and different clinical presentations (Baptista A, 2015). Due to this variable phenotype, the disease is still largely underdiagnosed. Therefore, the reports of a prevalence of ~1 per 40,000 / 100,000 persons in the general population are probably an underestimation (Terryn W, 2013). Previous screening studies for FD in high risk populations (left ventricular hypertrophy) report much higher frequencies, highlighting the need of including this disease among the differential diagnoses of left ventricular hypertrophy (LVH) of unexplained origin (Terryn W, 2012; Baptista A, 2015).

Left ventricular hypertrophy (LVH), detected both by imaging techniques (echocardiography, MRI) and by electrocardiography (ECG) is the predominant cardiac finding in Fabry patients (Linhart A, 2006). In a cross sectional study of untreated FD patients, half of the men and one third of the women were classified as having LVH (defined as LVMi of >51 g/m2.7 for males and >48 g/m2.7 for females) (Kampmann C, 2008). In screening studies in patients with LVH, the prevalence of FD is higher, including reports of a prevalence of up to 12% (Terryn W, 2012). Considering that enzyme replacement therapy (ERT) has been shown to significantly reduce left ventricular mass and wall thickness, an early diagnosis and treatment of these patients has the potential to modify the natural course of the disease and reduce morbidity and mortality. In addition, it offers the important possibility to diagnose family members in an earlier stage of the disease.

In FD, myocardial hypertrophy is known to be progressive over time and occurs earlier in men than in women. In female heterozygotes, suggested random X chromosome inactivation and the inability of the cells expressing the wild type allele to cross correct the metabolic defects lead to symptoms that are similar to those in hemizygous males (Linhard A, 2006). Due to the heterozygous status in female patients, diagnosis is much more difficult with direct genetic analysis representing the gold standard. Cardiovascular involvement substantially contributes to disease-related morbidity and mortality in FD. Over the past decade, several studies have suggested that FD can present regularly in patients with an echocardiographic phenotype of hypertrophic cardiomyopathy (HCM), defined by the presence of LVH in the absence of abnormal loading conditions such as arterial hypertension (AHT) or aortic valve abnormalities. It was supposed that these abnormal loading conditions generally explained LVH and therefore these patients were excluded in screening studies for FD so far. As a considerable part of the Fabry population has AHT and most of the patients with LVH followed by cardiologist in everyday practice have hypertension or valvular disease, a screening for FD in patients with LVH should include patients with hypertension and valvular disease, as will be the case in this current proposal. Establishing the cause of left ventricular hypertrophy (LVH) is a common challenge in clinical practice, given its high prevalence and the variety of diseases it may be associated with. This is particularly relevant from the clinical standpoint because of the therapeutic implications regarding the differential diagnoses. In this project we aim to assess the prevalence of FD in the Würzburg cohort of patients with LVH presenting over the last years. The results of this project will not only contribute to give the proper diagnosis and treatment to so far unidentified Fabry patients, but is also anticipated to help highlighting the relevance of considering FD as a possible cause of LVH in general clinical practice.

Primary study objective:

To identify FD patients in the Würzburg Cohort of patients with LVH of otherwise unexplained origin.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Written informed consent
* Preliminary diagnosis of hypertrophic non-obstructive cardiomyopathy

Exclusion Criteria:

* Severe outflow tract obstruction
* Positive genetic testing for sarcomeric HCM or other hereditary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Alpha Galactosidase level | 1 day (Once after inclusion & informed consent)
  A blood sample will be taken to determine alpha-galactosidase level. If alpha-galactosidase level is low, FD specific genetic testing is advised (outside this study in the regular clinical routine).
Lyso-GB3 level | 1 day (Once after inclusion & informed consent)
  A blood sample will be taken to determine alpha-galactosidase level. If LysoGb3-level is high, FD specific genetic testing is advised (outside this study in the regular clinical routine).
Genetic testing | 1 day (Once after inclusion & informed consent)
  Optional testing of fabry specific GLA-gene

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doheny D, Srinivasan R, Pagant S, Chen B, Yasuda M, Desnick RJ. Fabry Disease: prevalence of affected males and heterozygotes with pathogenic GLA mutations identified by screening renal, cardiac and stroke clinics, 1995-2017. J Med Genet. 2018 Apr;55(4):261-268. doi: 10.1136/jmedgenet-2017-105080. Epub 2018 Jan 12. PMID 29330335
- [Background] Kim WS, Kim HS, Shin J, Park JC, Yoo HW, Takenaka T, Tei C. Prevalence of Fabry Disease in Korean Men with Left Ventricular Hypertrophy. J Korean Med Sci. 2019 Feb 15;34(7):e63. doi: 10.3346/jkms.2019.34.e63. eCollection 2019 Feb 25. PMID 30804731
- [Derived] Lau K, Sokalski V, Lorenz L, Fette G, Sommer C, Uceyler N, Wanner C, Nordbeck P. Automated electronic health record-based screening for Fabry disease in unexplained left ventricular hypertrophy (FAPREV-HCM). Open Heart. 2025 Jan 11;12(1):e003116. doi: 10.1136/openhrt-2024-003116. PMID 39800432